CLINICAL TRIAL: NCT01429038
Title: Infusion of Third-party Mesenchymal Stem Cells After Renal or Liver Transplantation. A Phase I-II, Open-label, Clinical Study
Brief Title: Mesenchymal Stem Cells After Renal or Liver Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Yves Beguin, Prof, University of Liege
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJT1106P1
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Liver Failure; Kidney Failure
Keywords: end-stage; liver diseases; cirrhosis; cancer; fulminant hepatic failure; metabolic hepatic diseases; congenital hepatic diseases; renal diseases
MeSH Terms: conditions — Liver Failure; Renal Insufficiency; Liver Diseases; Fibrosis; Neoplasms; Liver Failure, Acute; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MSC Liver Transplantation (Experimental): Patients undergoing a first liver transplantation. Beside receiving standard liver tranplantation care (antibacterial and viral prophylactic treatments as well as a standard immunosuppressive regime i.e. tacrolimus, mycophenolate mofetil and steroids), patients will be infused with 1,5-3,0 10E6 MSC/kg on postoperative day 3+/-2
  Interventions: Biological: Mesenchymal Stem Cells
- MSC Kidney Transplantation (Experimental): Patients undergoing a first kidney transplantation. Beside receiving standard kidney tranplantation care (antibacterial and viral prophylactic treatments as well as a standard immunosuppressive regime i.e. tacrolimus, mycophenolate mofetil and steroids associated with ant-IL-2 antibodies), patients will be infused with 1,5-3,0 10E6 MSC/kg on postoperative day 3+/-2.
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — Third party MSC 1,5-3,010E6/kg. No HLA matching between MSC donor and the recipient or the liver/kidney donor. One infusion at day 3+/-2.
  Other Names: MSC

SUMMARY:
The immune system of a patient can attack the liver or the kidney received from a donor (organ rejection). This can be prevented by treating these patients long-life with immunosuppressive drugs. Unfortunately, these drugs lead to numerous side effects and fail to prevent the rejection occurring months later after the transplantation (chronic rejection). Recently, it has been shown that a particular type of cells present in the bone marrow, namely Mesenchymal Stem Cells (MSC), when injected to a patient, suppress its immune system and increase success rates of blood cells transplantation. This outcome opens doors to investigate the potential of these cells to provide a valuable tool for improving solid organ transplantation without the need of high concentration of immunosuppressive drugs. The present project aims at evaluating the safety and tolerability of MSC administration after liver or kidney transplantation.

DETAILED DESCRIPTION:
The present project aims at evaluating the safety and tolerability of third party MSC administration after liver or kidney organ transplantation. Ten patients undergoing liver transplantation and 10 patients undergoing kidney transplantation will be included in the experimental arm to receive a single infusion of MSC. The outcome of each of these 2 subgroups will be compared with that of similar control patients undergoing liver or kidney transplantation but who will not receive MSC.

Liver and kidney transplanted patients will receive standard immunosuppressive therapy, TAC-MMF-steroïds and TAC-MMF-steroïds plus an IL-2-R antibody respectively. Patients enrolled in the experimental arms will be infused with a single dose of 1,5-3,0 10E6 MSC/kg, 3(+/-2) days after the transplantation.

Weaning of immunosuppression will be attempted from month 6 in liver transplant patients who did not present a rejection episode and show normal graft function and graft biopsy.

Kidney transplant patients will continue standard immunosuppressive therapy indefinitely.

Male or female (>18 years) individuals unrelated to the recipient or the graft donor will be MSC donors. MSC donors need to fulfill generally accepted criteria for allogeneic HSC donation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 75 years of age, who will undergo first Kidney Transplantation or whole Liver Transplantation from a cadaveric or donation after cardiac death (DCD) organ donor;
* Fertile female patients must use a reliable contraception method;
* Informed consent given by patient or his/next of kin if the patient is unable to give informed consent, for the complete (MSC + follow-up) or partial(no MSC + follow-up) study;
* Successful liver/kidney transplantation, demonstration of organ function (improvement of INR in liver recipients and of creatinine in kidney recipients at 24-36h) and normal graft vasculature at Doppler examination.

Exclusion Criteria:

* Past history of malignant disease, with the exception of hepatocarcinoma within the Milan criteria for the Liver Transplantation patients;
* Active uncontrolled infection;
* HIV or HCV positive;
* EBV-negative;
* Retransplantation;
* Combined transplantation;
* Living related transplantation or split liver transplantation;
* Autoimmune disease or expected impossibility to wean immunosuppression (Liver Transplantation) or corticosteroids (Kidney Transplantation);
* Endotracheal intubation;
* Postoperative cardiovascular instability, active hemorrhage, or any other serious clinical complication between transplantation and evaluation for suitability for MSC infusion;
* For Kidney Transplantation: panel reactive antibodies (PRA) >50%.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Infusional toxicity | Within 24 hours of infusion
  Incidence, timing and severity of any clinical complication related to MSC infusion, including pulmonary events or immune reactions.
Incidence of infections (bacterial, viral, fungal, parasitic) and cancers | Continuously over 2 years
  * Incidence, timing and severity of any infection (bacterial, viral, fungal, parasitic) (blood hemoculture, urine culture, PCR CMV, PCR BK virus at month 1,2,3)
  * Incidence, timing and severity of malignant disease (Posttransplant lymphoproliferative disorder or other)

SECONDARY OUTCOMES:
Patient and graft survivals | Continuously over 2 years
Effects of MSC on graft function | over 1 year
  * Liver Transplantation: bilirubin, INR, transaminases, GGT, at day 7, months 1, 3, 6, 9, 12.
  * Kidney Transplanttaion: number of post transplant hemodialysis, creatinine at day 7, months 1, 3, 6, 9, 12.
Biopsy-proven (Banff classification) rejection rates | over 1 year
  At months 3, 6, 9, 12.
Feasibility and safety of weaning or decreasing immunosuppression | continuously over 2 years
  Decision points at months 3, 6, 9, 12.
Recipient's immune function | over 1 year
  To evaluate recipient's immune function (T cell blood populations (including T regs) by FACS, TREC quantification, Vβ repertoire diversity, pathogen-specific T cells, anti-organ donor HLA antibodies).
Anti-MSC donor HLA antibodies. | over 1 year
  To evaluate the potential development of anti-MSC donor HLA antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Beguin, MD, PhD, Principal Investigator — CHU-ULg
Locations (1):
- University Hospital Liege, Liège, Belgium

REFERENCES:
- [Derived] Detry O, Vandermeulen M, Delbouille MH, Somja J, Bletard N, Briquet A, Lechanteur C, Giet O, Baudoux E, Hannon M, Baron F, Beguin Y. Infusion of mesenchymal stromal cells after deceased liver transplantation: A phase I-II, open-label, clinical study. J Hepatol. 2017 Jul;67(1):47-55. doi: 10.1016/j.jhep.2017.03.001. Epub 2017 Mar 9. PMID 28284916